CLINICAL TRIAL: NCT03223961
Title: A Randomized Trial Testing Early vs Late Onset of EPO Alfa Treatment in Lower Risk MDS With Non RBC Transfusion Dependent Anemia and Without Del 5q
Brief Title: A Trial Testing Early vs Late Onset of EPO Alfa Treatment in Lower Risk MDS
Acronym: EPO-PRETAR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GFM-EPO-PRETAR
Record Dates: First submitted 2017-07-11; First posted 2017-07-21 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Myelodysplastic Syndromes
Keywords: myelodysplastic syndrome; erythropoetin
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Epoetin Alfa

STUDY DESIGN:
Intervention Model Description: randomazed study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early onset arm (Experimental): Intervention: early onset of Eprex60000 IU/week , at patient inclusion
  Interventions: Drug: EPREX
- Delayed onset arm (Experimental): Intervention: late introduction of Eprex60000 IU/week, whenever the patient reaches the level chosen RBC transfusions (based on age, comorbidities, anticipated tolerance of anemia).
  Interventions: Drug: EPREX

INTERVENTIONS:
Drug: EPREX — 60 000 U/week for at least 12 weeks
  Other Names: Epoetin alfa

SUMMARY:
This is an open-label, randomized, multicenter, phase III study

Patients with baseline Hb comprised between 9 and 10.5g/dl will be randomized to receive EPO Alfa 60000 UI/week for at least 12 weeks:

* Either at diagnosis Or
* at the Hb threshold chosen for RBC transfusions (must be < 9g/dl)

DETAILED DESCRIPTION:
in this trial we will compare the early introduction of EPO alfa to the delayed introduction in lower risk MDS with non RBC transfusion dependent anemia.

At enrollment patients will be randomised in the 2 arms (early and delayed start of EPO alfa).

Treatment Regimen Epoetin alfa 60000 UI/week for at least 12 weeks

1. Early onset arm: early onset of EPO ALFA 60000 IU/week , at patient inclusion
2. Delayed onset arm: late introduction of EPO ALFA 60000 IU/week, whenever the patient reaches the level chosen RBC transfusions (based on age, comorbidities, anticipated tolerance of anemia).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. MDS according to WHO 2016 criteria, with low or int 1 classical IPSS
3. Non-RBC transfusion dependent anemia
4. Hb level between 9 and 10.5g/dl (at the center's lab)
5. Hb level should be at least 1g/dl higher than the Hb threshold chosen to start RBC transfusions based on age, comorbidities and predicted clinical tolerance of anemia (this transfusion threshold should be chosen between 8 and 9g/dl)
6. Serum EPO level <500U/l
7. No other cause of anemia (including iron deficiency, vitamin B12 or B9 deficiency, hemolysis, hypothyroidism….)
8. Performance status <=2

Exclusion Criteria:

1. Higher risk MDS (IPSS intermediate-2 or high)
2. Del 5q
3. Baseline Hemoglobin level > 10.5 g/dl or <9g/dl
4. Transfusion threshold (based on age , comorbidities…) >9g/dl
5. Transfusion threshold less than 1 g/dl below baseline Hb level
6. RBC transfusion dependence. Patients may have received only one transfusion series for MDS prior to inclusion
7. CMML , if >10 % BM blasts or WBC>13.000/mm3
8. Uncontrolled hypertension
9. Uncontrolled cardiovascular disease including angina pectoris or cardiac failure
10. Renal failure: Creatinine clearance<40ml/min (using MDRD formula)
11. Pregnancy (positive bettaHCG) or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2018-03-26 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Time to RBC transfusion dependence in non RBC transfusion dependent lower risk MDS patients with anemia with early (at inclusion of the patient) versus delayed onset,( at the threshold chosen for RBC transfusion) of EPO ALFA | 12 weeks
  RBC transfusion dependence will be defined by requirement of at least transfusions of 2 PRBC within an interval of less than 8 weeks, given for Hb <8g/dl or <9g/dl according to comorbidities and in the absence of other cause of anemia (bleeding, surgery…), taking into account only transfusions given at least 12 weeks after onset of treatment with EPO ALFA.

SECONDARY OUTCOMES:
Erythroid response (according to IWG 2006 criteria) | 12 weeks
  Erythroid response (according to IWG 2006 criteria) after 12 weeks of EPO ALFA treatment
response duration to EPO ALFA | 4 years
  response duration to EPO ALFA measured from the date of enrollment until failure
Overall survival | 4 years
  Overall survival measured from the date of enrollment to death or the date of last contact

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Park, Prof, Principal Investigator — University Hospital, Grenoble
Locations (39):
- France (39):
  - Chu Amiens, Amiens
  - CH Angers, Angers
  - CH Avignon, Avignon
  - Centre Hospitalier de La Cote Basque, Bayonne
  - Hopital Nord Franche-Comté, Belfort
  - CHU de Besançon, Besançon
  - Hopital Avicenne, Bobigny
  - Hôpital Morvan, Brest
  - CHU de Caen, Caen
  - CH de Sevigné, Cesson
  - CH de Cholet, Cholet
  - CHU Estaing, Clermont-Ferrand
  - CHSF Gilles de Corbeil, Corbeil-Essonnes
  - Hôpital Henri-Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - Centre Hospitalier du Mans, Le Mans
  - Clinique Victor Hugo, Le Mans
  - Hopital Saint-Vincent de Paul, Lille
  - CHRU Limoges, Limoges
  - Centre Hospitalier Lyon Sud, Lyon
  - IPC, Marseille
  - Centre Hospitalier du Mont de Marsan, Mont-de-Marsan
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - Hopital St Louis T4, Paris
  - Centre Hospitalier Joffre-Perpignan, Perpignan
  - Sophie Dimicoli-Salazar, Pessac
  - CH de Périgueux, Périgueux
  - CHU de Poitiers, Poitiers
  - CHR d'Annecy, Pringy
  - CHRU de Reims, Reims
  - CHU Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - CH Saint Nazaire, Saint-Nazaire
  - Centre Hospitalier Universitaire de STRASBOURG, Strasbourg
  - IUCT Oncopole, Toulouse
  - CH de Troyes, Troyes
  - CH Valence, Valence
  - CHU Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Undecided